CLINICAL TRIAL: NCT02856737
Title: Reducing Delirium in the Surgical Intensive Care Unit Through the Use of Eye Masks and Earplugs
Brief Title: Reducing Delirium in the Surgical Intensive Care Unit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: inadequate personel
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Stephanie Talutis, Fellow in the Study of Quality and Patient Safety, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SICU Delirium
Record Dates: First submitted 2016-08-01; First posted 2016-08-05 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Ear Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Earplugs and eye masks (to be used concurrently) (Experimental): Group will include patients consented to the use of earplugs and eye masks. Patients will participate in the intervention nightly
  Interventions: Other: eye masks and earplugs

INTERVENTIONS:
Other: eye masks and earplugs — Materials similar to those offered on long commercial flights

SUMMARY:
Delirium is an acute disturbance in mental abilities and confusion that affects many patient in the hospital and is caused by multiple factors including and altered sleep/wake cycles and multiple sedating medications. Patients in the ICU are particularly susceptible to developing delirium due to increased noise levels and metabolic derangements.

Numerous studies have shown that delirium can be associated with many negative outcomes, including longer hospital length of stay, increased time on a ventilator, higher mortality rates, and greater long-term cognitive dysfunction. There are a series of non-pharmacological interventions that have been shown to reduce delirium especially in intensive care units. These include noise reduction, frequent reorientation, reducing unnecessary stimulation at night, and grouping patient care procedures.

The aim of this study is to evaluate the benefits of eye masks and earplugs (used concurrently) on reducing delirium and to assess for associated outcomes such as length of stay, use of sedating medications, morbidity, and mortality. The benefits of this are to improve sleep quality, and this intervention has been associated with a reduction in the risk of delirium.

DETAILED DESCRIPTION:
Delirium is an acute disturbance in mental abilities and confusion that affects many patient in the hospital and is caused by multiple factors including and altered sleep/wake cycles and multiple sedating medications. Patients in the ICU are particularly susceptible to developing delirium due to increased noise levels and metabolic derangements.

Numerous studies have shown that delirium can be associated with many negative outcomes, including longer hospital length of stay, increased time on a ventilator, higher mortality rates, and greater long-term cognitive dysfunction. There are a series of non-pharmacological interventions that have been shown to reduce delirium especially in intensive care units. These include noise reduction, frequent reorientation, reducing unnecessary stimulation at night, and grouping patient care procedures.

The aim of this study is to evaluate the benefits of eye masks and earplugs on reducing delirium and to assess for associated outcomes such as length of stay, use of sedating medications, morbidity, and mortality. The benefits of this are to improve sleep quality, and this intervention has been associated with a reduction in the risk of delirium.

Detailed Description: Patients eligible for this study will include patients admitted to either the Surgical ICU (SICU) or stepdown unit, under the care of the SICU care team, beginning on 8/1/16. Consent will be obtained from patients or their family members by study personnel. Data that will be collected include diagnosis on admission, any surgeries performed and their respective dates, length of stay in the SICU and step-down unit, use of sedating medication, and the Confusion Assessment Method (CAM) results. Subjects will also be asked to fill out 2 separate questionnaires about the quality of their sleep. The first questionnaire will be administered on enrollment and the second questionnaire will be administered upon discharge from the SICU. The rates of compliance of the use of earplugs and eye masks will also be assessed by means of a calendar checklist to be displayed at the patient's bedside.

These outcomes will be compared to those of a historical control group not undergoing such interventions. The investigators aim to enroll 100 subjects and have a control group of another 100 patients retrospectively selected from matched patients over the previous year (8/1/15 - 8/1/16), before implementation of such interventions. The remainder of patient data will be collected by means of a retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patient spending more than or equal to 24 hours in the SICU or stepdown unit

Exclusion Criteria:

* Known pre-existing history of sleep pathology, severe visual or hearing impairment
* History of cognitive dysfunction (dementia, traumatic brain injury, stroke or hepatic encephalopathy, or intellectual disability)
* Admitted in delirious state
* Facial trauma involving orbits or auditory canals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Delirium | for the duration of a patient's hospital stay (1 day - 1 year)
  Daily assessment of delirium documented in the patient's chart
Length of stay | for the duration of a patient's hospital stay (1 day - 1 year)
Sedative use | for the duration of a patient's hospital stay (1 day - 1 year)
  quantification of sedating medications used during a patient's hospital stay
CAM-ICU | for the duration of a patient's hospital stay (1 day - 1 year)
  documentation of the CAM-ICU scoring system for delirium on a daily basis in patient's chart

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie D Talutis, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNicoll L, Pisani MA, Zhang Y, Ely EW, Siegel MD, Inouye SK. Delirium in the intensive care unit: occurrence and clinical course in older patients. J Am Geriatr Soc. 2003 May;51(5):591-8. doi: 10.1034/j.1600-0579.2003.00201.x. PMID 12752832
- [Background] Pandharipande PP, Girard TD, Ely EW. Long-term cognitive impairment after critical illness. N Engl J Med. 2014 Jan 9;370(2):185-6. doi: 10.1056/NEJMc1313886. No abstract available. PMID 24401069
- [Background] Rivosecchi RM, Kane-Gill SL, Svec S, Campbell S, Smithburger PL. The implementation of a nonpharmacologic protocol to prevent intensive care delirium. J Crit Care. 2016 Feb;31(1):206-11. doi: 10.1016/j.jcrc.2015.09.031. Epub 2015 Oct 17. PMID 26596509
- [Background] Patel J, Baldwin J, Bunting P, Laha S. The effect of a multicomponent multidisciplinary bundle of interventions on sleep and delirium in medical and surgical intensive care patients. Anaesthesia. 2014 Jun;69(6):540-9. doi: 10.1111/anae.12638. PMID 24813132
- [Background] Huang HW, Zheng BL, Jiang L, Lin ZT, Zhang GB, Shen L, Xi XM. Effect of oral melatonin and wearing earplugs and eye masks on nocturnal sleep in healthy subjects in a simulated intensive care unit environment: which might be a more promising strategy for ICU sleep deprivation? Crit Care. 2015 Mar 19;19(1):124. doi: 10.1186/s13054-015-0842-8. PMID 25887528
- [Background] Litton E, Carnegie V, Elliott R, Webb SA. The Efficacy of Earplugs as a Sleep Hygiene Strategy for Reducing Delirium in the ICU: A Systematic Review and Meta-Analysis. Crit Care Med. 2016 May;44(5):992-9. doi: 10.1097/CCM.0000000000001557. PMID 26741578
- [Background] Van Rompaey B, Elseviers MM, Van Drom W, Fromont V, Jorens PG. The effect of earplugs during the night on the onset of delirium and sleep perception: a randomized controlled trial in intensive care patients. Crit Care. 2012 May 4;16(3):R73. doi: 10.1186/cc11330. PMID 22559080